CLINICAL TRIAL: NCT06804538
Title: Interest of Sperm Insemination at 42 Hours Post hCG Compared to 36h in Intrauterine Insemination : a Randomized Controlled Trial. SYNcIU
Brief Title: Interest of Sperm Insemination at 42 Hours Post hCG Compared to 36h in Intrauterine Insemination
Acronym: SYNcIU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/24/0309
Record Dates: First submitted 2025-01-09; First posted 2025-02-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Infertility; Intrauterine Insemination (IUI)
Keywords: intrauterine insemination; infertility; sperm donation; timing; live birth
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group: insemination between 42 and 43 hours post hCG (Experimental): Patients in the experimental group will be stimulated by gonadotropins, ovulation will be blocked by a GnRH antagonist then triggered by hCG allowing IU to occur between 42 and 43 hours post hCG. These treatments are similar to the control group. Only the timing of the IUI compared to the timing of ovulation triggering is different
  Interventions: Procedure: Insemination between 42 and 43 hours post hCG
- Control group: insemination between 36 and 37 hours post hCG (Active Comparator): In the comparison group, patients will be stimulated with gonadotropin and GnRH antagonist whose ovulation will be triggered and for which intrauterine insemination will be carried out between 36 and 37 hours post hCG (as it is already the case in clinical practice).
  Interventions: Procedure: Insemination between 36 and 37 hours post hCG

INTERVENTIONS:
Procedure: Insemination between 42 and 43 hours post hCG — Patients will be stimulated by gonadotropins, ovulation will be blocked by a GnRH antagonist then triggered by hCG allowing IU to occur between 42 and 43 hours post hCG
  Arms: Experimental group: insemination between 42 and 43 hours post hCG
Procedure: Insemination between 36 and 37 hours post hCG — Patients will be stimulated with gonadotropin and GnRH antagonist whose ovulation will be triggered and for which intrauterine insemination will be carried out between 36 and 37 hours post hCG
  Arms: Control group: insemination between 36 and 37 hours post hCG

SUMMARY:
Intrauterine insemination (IUI) is a common therapeutic option to treate infertility. Typically performed 36 hours post-hCG injection to trigger ovulation. However, research suggests delaying IUI to 42 hours post-hCG may improve egg quality and sperm synchronization for fertilization, leading to higher pregnancy rates. A proposed superiority study aims to compare IUI timing at 36 hours versus 42 hours post-hCG injection to evaluate its impact on live birth rates. The primary objective is to assess the effectiveness (live birth rates) of IUI at two different post-hCG timing intervals (42-43 hours vs 36-37 hours).

DETAILED DESCRIPTION:
Infertility is a major problem affecting approximately 15% of couples worldwide, with a notable increase due to various factors such as advanced maternal age and unhealthy lifestyles. Intrauterine insemination (IUI) is a common treatment option that aims to increase the chances of conception. It is preceded by ovarian stimulation to promote the growth of the follicles. Traditionally, IUI is performed 36 hours after an hCG injection to trigger ovulation, but research suggests benefits to delaying it. Studies have shown that delaying IUI to 42 hours post-hCG could improve oocyte quality and sperm synchronization for fertilization. Randomized clinical trials have shown higher pregnancy rates with delayed UTIs to 42 hours. We therefore propose a superiority study to compare IU at 36 hours and 42 hours post-hCG, taking into account the origin of the sperm used. This study will be the first to evaluate the effect of hCG-IU delay on live birth rates. In all centers, inseminations will be carried out according to the usual procedure. Patients in the experimental group will be stimulated by gonadotropins, ovulation will be blocked by a GnRH antagonist then triggered by hCG allowing IU to occur between 42 and 43 hours post hCG. These treatments are similar to the control group. Only the timing of the IUI compared to the timing of ovulation triggering is different. In the comparison group, ovulation will be triggered in order to carry out intrauterine insemination between 36 and 37 hours post hCG (as is already the case in clinical practice). Blinding is not possible for this study. On the other hand, the different endpoints will be evaluated without the randomization group being blinded by the evaluating gynaecologists. The monitoring of included patients is similar to the care pathway. The follow-up data (pregnancy test, pregnancy ultrasound, progress of the birth) will be carried out in the same way as the care (for which these data are necessarily collected)

ELIGIBILITY:
Inclusion Criteria:

* Single unmarried woman or heterosexual or homosexual couple in which the woman wishing to carry the pregnancy is aged 18 to 43 and the spouse is aged 18 to 60 at the time of inclusion
* 2 permeable tubes for the woman receiving the insemination
* Spouse's sperm (Number of inseminable sperm ≥ 1 million in prior survival migration test) or sperm donation
* 1st or 2nd intrauterine insemination for this child project
* Ovarian stimulation by gonadotropin with GnRH antagonist (introduced on a fixed day or according to the follicular size criterion of the center)
* Luteal phase support with a progestin until at least the pregnancy test
* Affiliation or beneficiary of a social security scheme or equivalent for both partners of the couple if applicable
* Free and informed consent signed by the unmarried woman or both members of the couple
* Couples and unmarried women meeting the conditions for access to PMA according to the French bioethics law

Exclusion Criteria:

* Endometriosis stage III or IV
* History of ectopic pregnancy
* ≥ 3 spontaneous miscarriages
* Single woman or couple where one of the two partners (or both) is (are) under the protection of justice, under guardianship or under curatorship
* Single woman or couple who have already participated in the study once
* Single woman or couple participating in another interventional clinical study

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Single unmarried woman or heterosexual or homosexual couple in which the woman wishing to carry the pregnancy is aged 18 to 43 and the spouse is aged 18 to 60 at the time of inclusion because the study concerns intrauterine insemination
Enrollment: 692 (Estimated)
Dates: Start 2025-09-09 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Delivery rate after 22 weeks of pregnancy with at least one live birth per woman | the day of delivery
  The live birth rate is the most relevant clinical criterion for judging the effectiveness (success) of the IUI attempt. This criterion will be evaluated according to the usual procedures of the centers via the obligatory collection of post-ART childbirth data and transmission in a regulatory manner to the Biomedicine Agency.

SECONDARY OUTCOMES:
Biochemical pregnancy rate | The day of the pregnancy test: 15 days after insemination (T0)
  Number of β-hCG >100 IU/l
Clinical pregnancy rate | During ultrasound realised at 6 weeks' amenorrhea (SA)
  Presence of at least one intrauterine gestational sac with fetal heart activity.
Spontaneous miscarriage rate | The day of delivery before 22 weeks of pregnancy
  Number of pregnancies terminated before 22 weeks of pregnancy/number of biochemical pregnancies

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Bordeaux, Bordeaux
  - CHU La Réunion, La Réunion
  - CHU Poitiers, Poitiers
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No